CLINICAL TRIAL: NCT05039814
Title: Prediction of Postoperative Acute Kidney Injury in Patients With Acute Type A Aortic Dissection Using Cystatin C
Status: Completed | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: 81500367
Record Dates: First submitted 2021-09-01; First posted 2021-09-10 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2021-08

CONDITIONS: Aortic Dissection; Acute Kidney Injury
MeSH Terms: conditions — Aortic Dissection; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- AKI: patients suffered postoperative acute kidney injury
  Interventions: Other: postoperative acute kidney injury
- Non-AKI: patients did not suffer postoperative acute kidney injury
  Interventions: Other: none postoperative acute kidney injury

INTERVENTIONS:
Other: postoperative acute kidney injury — patients suffered postoperative acute kidney injury
  Groups: AKI
Other: none postoperative acute kidney injury — patients did not suffered postoperative acute kidney injury
  Groups: Non-AKI

SUMMARY:
The research aimed to predict postoperative acute kidney injury in patients with acute type A aortic dissection preliminarily by exploring the correlation of preoperative cystatin C level and incidence of postoperative acute kidney injury and combining with relevant risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old
2. Acute type A aortic dissection diagnosed by CT angiography

Exclusion Criteria:

1. History of chronic kidney disease
2. History of cardiovascular operation
3. Pregnancy status

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients sufferred acute type A aortic dissection
Sampling Method: Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
postoperative acute kidney injury | From date of operation until the date of acute kidney injury or date of death from any cause, whichever came first, assessed up to 30 days.
  YES; NO

CONTACTS AND LOCATIONS:
Overall Officials: Xin Zhao, Principal Investigator — Department of cardiac surgery, Qilu Hospital, Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided